CLINICAL TRIAL: NCT00818259
Title: A Multicenter, Open-Label, 5-Part Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Aprepitant and Fosaprepitant Dimeglumine in Pediatric Patients Receiving Emetogenic Chemotherapy
Brief Title: A Study of MK-0869 (Aprepitant) and MK-0517 (Fosaprepitant) in Pediatric Participants Receiving Chemotherapy (MK-0869-134)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated early prior to completing targeted enrollment of participants <6 months of age due to recruitment challenges.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0869-134; 2009_501 (Other: Telerx Study Identifier)
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-08

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Aprepitant; fosaprepitant; Ondansetron; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Part IA-fosaprepitant 115 mg/aprepitant (Experimental): Day 1, fosaprepitant intravenous (IV) at a dose of 115 mg and Days 2 and 3, aprepitant 80 mg orally (PO), prior to chemotherapy for participants from 12 to 17 years of age. Participants also receive ondansetron IV as per local standard of care, with or without dexamethasone IV.
  Interventions: Drug: Experimental: aprepitant; Drug: Experimental: fosaprepitant; Drug: Ondansetron; Drug: Dexamethasone
- Part IB-fosaprepitant 150 mg (Experimental): Day 1, fosaprepitant, IV at a dose of 150 mg, prior to chemotherapy for participants 12 to 17 years of age. Participants also receive ondansetron IV as per local standard of care, with or without dexamethasone IV.
  Interventions: Drug: Experimental: fosaprepitant; Drug: Ondansetron; Drug: Dexamethasone
- Part IIA-aprepitant 80 mg equiv. (Experimental): Day 1, aprepitant PO prior to chemotherapy at the dosing regimens listed for the following age ranges: 6 months to <12 years of age - 47 mg/m^2; 4 months to <6 months of age - 2.0 mg/kg; 1 month to <4 months of age - 1.0 mg/kg; birth to <1 month of age - 0.5 mg/kg. Participants also receive ondansetron IV as per local standard of care, with or without dexamethasone IV.
  Interventions: Drug: Experimental: aprepitant; Drug: Ondansetron; Drug: Dexamethasone
- Part IIB-aprepitant 125 mg equiv. (Experimental): Day 1, aprepitant PO prior to chemotherapy at the dosing regimens listed for the following age ranges: 2 years to <12 years of age - 74 mg/m^2; 6 months to <2 years of age - 1.3 mg/kg; 4 months to <6 months of age - 3.0 mg/kg; 1 month to <4 months of age - 1.5 mg/kg; birth to <1 month of age - 0.75 mg/kg. Participants also receive ondansetron IV as per local standard of care, with or without dexamethasone IV.
  Interventions: Drug: Experimental: aprepitant; Drug: Ondansetron; Drug: Dexamethasone
- Part III-ondansetron (Active Comparator): Ondansetron administered IV per local standard of care on Days 1, 2, and 3 prior to chemotherapy for participants from birth to <12 years of age. The use of IV dexamethasone is optional with the exception of the birth to one year old cohort.
  Interventions: Drug: Comparator: ondansetron; Drug: Dexamethasone
- Part IV-aprepitant regimen (Experimental): Day 1, aprepitant, PO, prior to chemotherapy at the dosing regimens listed for the following age ranges: 4 months to <12 years of age - 3.0 mg/kg; 1 month to <4 months of age - 1.5 mg/kg; Birth to <1 month of age - 0.75 mg/kg; Days 2 and 3, aprepitant, PO, prior to chemotherapy at the dosing regimens listed for the following age ranges: 4 months to <12 years of age - 2.0 mg/kg; 1 month to <4 months of age - 1.0 mg/kg; Birth to <1 month of age - 0.5 mg/kg. Participants also receive ondansetron IV as per local standard of care. The use of dexamethasone IV is optional with the exception of the birth to one year old cohort.
  Interventions: Drug: Experimental: aprepitant; Drug: Ondansetron; Drug: Dexamethasone
- Part V-fosaprepitant regimen (Experimental): Day 1, fosaprepitant, IV at a dose of 3 mg/kg prior to chemotherapy for participants 6 months to <12 years of age. Participants also receive ondansetron IV as per local standard of care, with or without dexamethasone IV.
  Interventions: Drug: Experimental: fosaprepitant; Drug: Ondansetron; Drug: Dexamethasone

INTERVENTIONS:
Drug: Experimental: aprepitant — aprepitant powder for suspension, 125 mg/sachet, PO
  Other Names: Emend; MK-0869
  Arms: Part IA-fosaprepitant 115 mg/aprepitant; Part IIA-aprepitant 80 mg equiv.; Part IIB-aprepitant 125 mg equiv.; Part IV-aprepitant regimen
Drug: Experimental: fosaprepitant — fosaprepitant lyophilized powder for suspension, 115 mg/vial or 150 mg/vial, IV
  Other Names: Emend injection; Fosaprepitant Dimeglumine; MK-0517
  Arms: Part IA-fosaprepitant 115 mg/aprepitant; Part IB-fosaprepitant 150 mg; Part V-fosaprepitant regimen
Drug: Comparator: ondansetron — ondansetron solution for infusion, IV, administered per local standard of care
  Other Names: Zofran
  Arms: Part III-ondansetron
Drug: Ondansetron — ondansetron solution for infusion, IV, administered per local standard of care
  Arms: Part IA-fosaprepitant 115 mg/aprepitant; Part IB-fosaprepitant 150 mg; Part IIA-aprepitant 80 mg equiv.; Part IIB-aprepitant 125 mg equiv.; Part IV-aprepitant regimen; Part V-fosaprepitant regimen
Drug: Dexamethasone — dexamethasone solution for infusion, IV, administered per local standard of care

SUMMARY:
This study will determine the appropriate dosing regimen of aprepitant and fosaprepitant for the prevention of chemotherapy-induced nausea and vomiting in pediatric participants from 0 months to 17 years of age.

DETAILED DESCRIPTION:
Fosaprepitant is a prodrug for aprepitant and is rapidly converted to aprepitant after intravenous administration; the pharmacological effect of fosaprepitant is attributed to aprepitant. The birth to one year old cohort will be initiated in Parts III and IV upon completion of Part II (Steps A and B) in participants <6 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Is 0 (at least 37 weeks gestation) to 17 years of age
* Is scheduled to receive moderately to highly nausea-inducing chemotherapy or participant did not tolerate a previous chemotherapy regimen that is planned to be repeated
* Is expected to receive ondansetron
* Female participants who have begun menstruating must have a negative pregnancy test
* Weighs ≥3.0 kg if <6 months of age, ≥6.0 kg if >6 months of age, and ≥7.5 kg if > 2 years of age
* Has a pre-existing venous catheter

Exclusion Criteria:

* Uses any illicit drugs or abuses alcohol
* Is pregnant or breast feeding
* Has a symptomatic central nervous system (CNS) tumor
* Has an infection or other uncontrolled disease other than cancer
* Has known history of heart QT wave prolongation

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2009-02-05 (Actual); Primary Completion 2014-01-20 (Actual); Study Completion 2014-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Kang HJ, Loftus S, Taylor A, DiCristina C, Green S, Zwaan CM. Aprepitant for the prevention of chemotherapy-induced nausea and vomiting in children: a randomised, double-blind, phase 3 trial. Lancet Oncol. 2015 Apr;16(4):385-94. doi: 10.1016/S1470-2045(15)70061-6. Epub 2015 Mar 12. PMID 25770814
- Available data/document: CSR Snyopsis — http://www.merck.com/clinical-trials/study.html?id=0869-134&kw=0869-134&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 92 unique participants who were enrolled and randomized in Parts I (n=23), II (n=39), III (n=19), IV (n=5) and V (n=6), 91 took part in this study. One participant randomized in Part IIB was discontinued prior to treatment.
Groups:
- Part IV-Additional Enrollers: Additional participants were enrolled in Part IV. Day 1, aprepitant, PO, prior to chemotherapy at the dosing regimens listed for the following age ranges: 4 months to <12 years of age - 3.0 mg/kg; 1 month to <4 months of age - 1.5 mg/kg; Birth to <1 month of age - 0.75 mg/kg; Days 2 and 3, aprepitant, PO, prior to chemotherapy at the dosing regimens listed for the following age ranges: 4 months to <12 years of age - 2.0 mg/kg; 1 month to <4 months of age - 1.0 mg/kg; Birth to <1 month of age - 0.5 mg/kg. Participants also receive ondansetron IV as per local standard of care. The use of dexamethasone IV is optional with the exception of the birth to one year old cohort.
- Part V-Additional Enrollers: Additional participants were enrolled in Part V. Day 1, fosaprepitant, IV at a dose of 3 mg/kg prior to chemotherapy for participants 6 months to <12 years of age. Participants also receive ondansetron IV as per local standard of care, with or without dexamethasone IV.
Period: Randomization
Arm/Group | Part IA-fosaprepitant 115 mg/Aprepitant | Part IB-fosaprepitant 150 mg | Part IIA-aprepitant 80 mg Equiv. | Part IIB-aprepitant 125 mg Equiv. | Part III-ondansetron | Part IV-aprepitant Regimen | Part IV-Additional Enrollers | Part V-fosaprepitant Regimen | Part V-Additional Enrollers
Started | 12 | 11 | 19 | 20 | 19 | 0 | 5 | 0 | 6
Completed | 12 | 11 | 19 | 20 | 19 | 0 | 5 | 0 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part I
Arm/Group | Part IA-fosaprepitant 115 mg/Aprepitant | Part IB-fosaprepitant 150 mg | Part IIA-aprepitant 80 mg Equiv. | Part IIB-aprepitant 125 mg Equiv. | Part III-ondansetron | Part IV-aprepitant Regimen | Part IV-Additional Enrollers | Part V-fosaprepitant Regimen | Part V-Additional Enrollers
Started | 12 (Newly enrolled participants) | 11 (Newly enrolled participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 11 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part II
Arm/Group | Part IA-fosaprepitant 115 mg/Aprepitant | Part IB-fosaprepitant 150 mg | Part IIA-aprepitant 80 mg Equiv. | Part IIB-aprepitant 125 mg Equiv. | Part III-ondansetron | Part IV-aprepitant Regimen | Part IV-Additional Enrollers | Part V-fosaprepitant Regimen | Part V-Additional Enrollers
Started | 0 | 0 | 19 (Newly enrolled participants) | 20 (Newly enrolled participants) | 0 | 0 | 0 | 0 | 0
Treated | 0 | 0 | 19 | 19 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 18 | 18 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Not Treated | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Part III
Arm/Group | Part IA-fosaprepitant 115 mg/Aprepitant | Part IB-fosaprepitant 150 mg | Part IIA-aprepitant 80 mg Equiv. | Part IIB-aprepitant 125 mg Equiv. | Part III-ondansetron | Part IV-aprepitant Regimen | Part IV-Additional Enrollers | Part V-fosaprepitant Regimen | Part V-Additional Enrollers
Started | 0 | 0 | 0 | 0 | 19 (Newly enrolled participants) | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 19 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part IV
Arm/Group | Part IA-fosaprepitant 115 mg/Aprepitant | Part IB-fosaprepitant 150 mg | Part IIA-aprepitant 80 mg Equiv. | Part IIB-aprepitant 125 mg Equiv. | Part III-ondansetron | Part IV-aprepitant Regimen | Part IV-Additional Enrollers | Part V-fosaprepitant Regimen | Part V-Additional Enrollers
Started | 0 | 0 | 0 | 0 | 0 | 15 (Participants continuing from Part III) | 5 (Newly enrolled participants) | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 14 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Part V
Arm/Group | Part IA-fosaprepitant 115 mg/Aprepitant | Part IB-fosaprepitant 150 mg | Part IIA-aprepitant 80 mg Equiv. | Part IIB-aprepitant 125 mg Equiv. | Part III-ondansetron | Part IV-aprepitant Regimen | Part IV-Additional Enrollers | Part V-fosaprepitant Regimen | Part V-Additional Enrollers
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 (Participants continuing from Part IV) | 6 (Newly enrolled participants)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: For analysis purposes, baseline (BL) data are presented by study part groups. The BL analysis population includes all unique enrolled participants in Parts I, II, III, IV and V. Part III participants who entered Parts IV and V are only counted in Part III; Part IV participants who entered Part V are only counted in Part IV.
Groups:
- Part IA-fosaprepitant 115 mg/Aprepitant: Day 1, fosaprepitant IV at a dose of 115 mg and Days 2 and 3, aprepitant 80 mg PO, prior to chemotherapy for participants from 12 to 17 years of age. Participants also receive ondansetron IV as per local standard of care, with or without dexamethasone IV.
- Total: Total of all reporting groups
Arm/Group | Part IA-fosaprepitant 115 mg/Aprepitant | Part IB-fosaprepitant 150 mg | Part IIA-aprepitant 80 mg Equiv. | Part IIB-aprepitant 125 mg Equiv. | Part III-ondansetron | Part IV-aprepitant Regimen | Part V-fosaprepitant Regimen | Total
Number analyzed (Participants) | 12 | 11 | 19 | 20 | 19 | 5 | 6 | 92
Age, Customized [Number; unit: Participants]
  6 months to <2 years | 0 | 0 | 5 | 6 | 6 | 1 | 1 | 19
  2 years to <6 years | 0 | 0 | 8 | 8 | 6 | 0 | 3 | 25
  6 years to <12 years | 0 | 0 | 6 | 6 | 7 | 4 | 2 | 25
  12 years to 17 years | 12 | 11 | 0 | 0 | 0 | 0 | 0 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 12 | 14 | 13 | 3 | 6 | 62
  Male | 5 | 4 | 7 | 6 | 6 | 2 | 0 | 30

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Time-Concentration Curve From 0 to 24 Hours (AUC 0-24hr) for Aprepitant
Description: AUC is a measure of the amount of aprepitant in the plasma. Fosaprepitant is a prodrug for aprepitant and is rapidly converted to aprepitant after IV administration. Blood samples for pharmacokinetic (PK) assessment were collected at the following time points: Part IA - Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 3, 4, 6, 8 and 24 hours (hr) post fosaprepitant dose; Part IB - Pre-dose and -0.75, -0.5, 0, 0.5, 1.5, 3, 4, 6, 8 and 24 hr post start of chemotherapy; Parts II and IV - Pre-dose and 1.5, 3, 4, 6, 8 and 24 hr post aprepitant dose; Part V - Pre-dose and -0.75, -0.5, 0, 1.5, 3, 4, 6, 8 and 24 hr post start of chemotherapy.
Time Frame: Up to 24 hours post fosaprepitant/aprepitant dose
Population: The population consisted of all participants who received at least one dose of fosaprepitant and/or aprepitant and were evaluable for this PK parameter. No PK assessements were performed on the Part III-ondansetron group; this group received no aprepitant.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Part IA-fosaprepitant 115 mg/Aprepitant | Part IB-fosaprepitant 150 mg | Part IIA-aprepitant 80 mg Equiv. | Part IIB-aprepitant 125 mg Equiv. | Part III-ondansetron | Part IV-aprepitant Regimen | Part V-fosaprepitant Regimen
Number analyzed (Participants) | 8 | 11 | 19 | 18 | 0 | 18 | 21
hr*ng/mL
  6 months to <2 years (n=0, 0, 5, 5, 0, 6, 6) | NA (NA) — Not assessed | NA (NA) — Not assessed | 20000 (7890) | 6310 (2040) |  | 21100 (11800) | 11700 (6980)
  2 years to <6 years (n=0, 0, 8, 7, 0, 6, 7) | NA (NA) — Not assessed | NA (NA) — Not assessed | 16400 (8080) | 23000 (8390) |  | 17300 (5060) | 18300 (11100)
  6 years to <12 years (n=0, 0, 6, 6, 0, 6, 8) | NA (NA) — Not assessed | NA (NA) — Not assessed | 16000 (4810) | 22000 (9440) |  | 24400 (15800) | 19500 (6720)
  12 years to 17 years (n=8, 11, 0, 0, 0, 0, 0) | 19500 (8010) | 30800 (7020) | NA (NA) — Not assessed | NA (NA) — Not assessed |  | NA (NA) — Not assessed | NA (NA) — Not assessed

2. Primary Outcome: Maximum Plasma Concentration (Cmax) for Aprepitant
Description: Cmax is a measure of the maximum amount of aprepitant in the plasma. Fosaprepitant is a prodrug for aprepitant and is rapidly converted to aprepitant after IV administration. Blood samples for PK assessment were collected at the following time points: Part IA - Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 3, 4, 6, 8 and 24 hr post fosaprepitant dose; Part IB - Pre-dose and -0.75, -0.5, 0, 0.5, 1.5, 3, 4, 6, 8, 24, 48 and 72 hr post start of chemotherapy; Parts II and IV - Pre-dose and 1.5, 3, 4, 6, 8, 24, 48 and 72 hr post aprepitant dose; Part V - Pre-dose and -0.75, -0.5, 0, 1.5, 3, 4, 6, 8, 24, 48 and 72 hr post start of chemotherapy.
Time Frame: Up to 72 hours post fosaprepitant/aprepitant dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part IA-fosaprepitant 115 mg/Aprepitant | Part IB-fosaprepitant 150 mg | Part IIA-aprepitant 80 mg Equiv. | Part IIB-aprepitant 125 mg Equiv. | Part III-ondansetron | Part IV-aprepitant Regimen | Part V-fosaprepitant Regimen
Number analyzed (Participants) | 12 | 11 | 19 | 18 | 0 | 19 | 22
ng/mL
  6 months to <2 years (n=0, 0, 5, 5, 0, 6, 7) | NA (NA) — Not assessed | NA (NA) — Not assessed | 1930 (1000) | 659 (107) |  | 1810 (925) | 1700 (636)
  2 years to <6 years (n=0, 0, 8, 7, 0, 6, 7) | NA (NA) — Not assessed | NA (NA) — Not assessed | 1300 (609) | 2100 (1170) |  | 1840 (933) | 2430 (1100)
  6 years to <12 years (n=0, 0, 6, 6, 0, 7, 8) | NA (NA) — Not assessed | NA (NA) — Not assessed | 1300 (275) | 1930 (873) |  | 1800 (1610) | 2850 (641)
  12 years to 17 years (n=12, 11, 0, 0, 0, 0, 0) | 3240 (1280) | 5870 (2770) | NA (NA) — Not assessed | NA (NA) — Not assessed |  | NA (NA) — Not assessed | NA (NA) — Not assessed

3. Primary Outcome: Time to Cmax (Tmax) for Aprepitant
Description: Tmax is a measure of the amount of time after dosing to when the maximum concentration of aprepitant was achieved. Fosaprepitant is a prodrug for aprepitant and is rapidly converted to aprepitant after IV administration. Blood samples for PK assessment were collected at the following time points: Part IA - Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 3, 4, 6, 8 and 24 hr post fosaprepitant dose; Part IB - Pre-dose and -0.75, -0.5, 0, 0.5, 1.5, 3, 4, 6, 8, 24, 48 and 72 hr post start of chemotherapy; Parts II and IV - Pre-dose and 1.5, 3, 4, 6, 8, 24, 48 and 72 hr post aprepitant dose; Part V - Pre-dose and -0.75, -0.5, 0, 1.5, 3, 4, 6, 8, 24, 48 and 72 hr post start of chemotherapy.
Time Frame: Up to 72 hours post fosaprepitant/aprepitant dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Part IA-fosaprepitant 115 mg/Aprepitant | Part IB-fosaprepitant 150 mg | Part IIA-aprepitant 80 mg Equiv. | Part IIB-aprepitant 125 mg Equiv. | Part III-ondansetron | Part IV-aprepitant Regimen | Part V-fosaprepitant Regimen
Number analyzed (Participants) | 12 | 11 | 19 | 18 | 0 | 19 | 22
hr
  6 months to <2 years (n=0, 0, 5, 5, 0, 6, 7) | NA (NA) — Not assessed | NA (NA) — Not assessed | 2.33 (1.16) | 3.45 (2.89) |  | 7.34 (8.28) | 1.13 (0.17)
  2 years to <6 years (n=0, 0, 8, 7, 0, 6, 7) | NA (NA) — Not assessed | NA (NA) — Not assessed | 3.78 (1.92) | 5.28 (1.97) |  | 4.92 (2.20) | 1.41 (0.83)
  6 years to <12 years (n=0, 0, 6, 6, 0, 7, 8) | NA (NA) — Not assessed | NA (NA) — Not assessed | 5.17 (1.83) | 3.08 (0.95) |  | 6.42 (7.84) | 1.07 (0.11)
  12 years to 17 years (n=12, 11, 0, 0, 0, 0, 0) | 0.41 (0.27) | 0.64 (0.30) | NA (NA) — Not assessed | NA (NA) — Not assessed |  | NA (NA) — Not assessed | NA (NA) — Not assessed

4. Primary Outcome: Apparent Terminal Half-life (t1/2) for Aprepitant
Description: t1/2 is the amount of time from dosing until half of the aprepitant was metabolized from the body. Fosaprepitant is a prodrug for aprepitant and is rapidly converted to aprepitant after IV administration. Blood samples for PK assessment were collected at the following time points: Part IA - Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 3, 4, 6, 8 and 24 hr post fosaprepitant dose; Part IB - Pre-dose and -0.75, -0.5, 0, 0.5, 1.5, 3, 4, 6, 8, 24, 48 and 72 hr post start of chemotherapy; Parts II and IV - Pre-dose and 1.5, 3, 4, 6, 8, 24, 48 and 72 hr post aprepitant dose; Part V - Pre-dose and -0.75, -0.5, 0, 1.5, 3, 4, 6, 8, 24, 48 and 72 hr post start of chemotherapy.
Time Frame: Up to 72 hours post fosaprepitant/aprepitant dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Part IA-fosaprepitant 115 mg/Aprepitant | Part IB-fosaprepitant 150 mg | Part IIA-aprepitant 80 mg Equiv. | Part IIB-aprepitant 125 mg Equiv. | Part III-ondansetron | Part IV-aprepitant Regimen | Part V-fosaprepitant Regimen
Number analyzed (Participants) | 6 | 11 | 16 | 13 | 0 | 12 | 21
hr
  6 months to <2 years (n=0, 0, 5, 3, 0, 3, 6) | NA (NA) — Not assessed | NA (NA) — Not assessed | 7.28 (1.47) | 8.09 (2.54) |  | 6.18 (4.12) | 7.71 (3.10)
  2 years to <6 years (n=0, 0, 6, 4, 0, 5, 7) | NA (NA) — Not assessed | NA (NA) — Not assessed | 8.27 (2.67) | 6.06 (3.03) |  | 9.21 (5.57) | 6.44 (2.35)
  6 years to <12 years (n=0, 0, 5, 6, 0, 4, 8) | NA (NA) — Not assessed | NA (NA) — Not assessed | 9.17 (4.00) | 6.89 (1.35) |  | 10.8 (4.27) | 8.76 (3.34)
  12 years to 17 years (n=6 11, 0, 0, 0, 0, 0) | 11.0 (4.42) | 22.2 (19.8) | NA (NA) — Not assessed | NA (NA) — Not assessed |  | NA (NA) — Not assessed | NA (NA) — Not assessed

5. Primary Outcome: Cmax for Fosaprepitant
Description: Cmax is a measure of the maximum amount of fosaprepitant in the plasma. Blood samples for PK assessment were collected at the following time points: Part IA - Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 3, 4, 6, 8 and 24 hr post fosaprepitant dose; Part V - Pre-dose and -0.75, -0.5, 0, 0.5, 1.5, 3, 4, 6, 8, 24, 48 and 72 hr post start of chemotherapy.
Time Frame: Up to 72 hours post fosaprepitant dose
Population: The population consisted of all participants who received at least one dose of fosaprepitant & were evaluable for this PK parameter. No PK analyses were performed on the Part 1A-fosaprepitant 115 mg/aprepitant group; blood samples from this group were not handled correctly. Part IIA, Part IIB, Part III & Part IV groups received no fosaprepitant.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part IA-fosaprepitant 115 mg/Aprepitant | Part IB-fosaprepitant 150 mg | Part IIA-aprepitant 80 mg Equiv. | Part IIB-aprepitant 125 mg Equiv. | Part III-ondansetron | Part IV-aprepitant Regimen | Part V-fosaprepitant Regimen
Number analyzed (Participants) | 0 | 11 | 0 | 0 | 0 | 0 | 23
ng/mL
  6 months to <2 years (n=0, 0, 0, 0, 0, 0, 7) |  | NA (NA) — Not assessed |  |  |  |  | 2756 (3364)
  2 years to <6 years (n=0, 0, 0, 0, 0, 0, 8) |  | NA (NA) — Not assessed |  |  |  |  | 3034 (1718)
  6 years to <12 years (n=0, 0, 0, 0, 0, 0, 8) |  | NA (NA) — Not assessed |  |  |  |  | 1654 (1995)
  12 years to 17 years (n=0, 11, 0, 0, 0, 0, 0) |  | 1310 (964) |  |  |  |  | NA (NA) — Not assessed

6. Primary Outcome: Tmax for Fosaprepitant
Description: Tmax is a measure of the amount of time after dosing to when the maximum concentration of fosaprepitant was achieved. Blood samples for PK assessment were collected at the following time points: Part IA - Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 3, 4, 6, 8 and 24 hr post fosaprepitant dose; Part V - Pre-dose and -0.75, -0.5, 0, 0.5, 1.5, 3, 4, 6, 8, 24, 48 and 72 hr post start of chemotherapy.
Time Frame: Up to 72 hours post fosaprepitant dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Part IA-fosaprepitant 115 mg/Aprepitant | Part IB-fosaprepitant 150 mg | Part IIA-aprepitant 80 mg Equiv. | Part IIB-aprepitant 125 mg Equiv. | Part III-ondansetron | Part IV-aprepitant Regimen | Part V-fosaprepitant Regimen
Number analyzed (Participants) | 0 | 11 | 0 | 0 | 0 | 0 | 22
hr
  6 months to <2 years (n=0, 0, 0, 0, 0, 0, 7) |  | NA (NA) — Not assessed |  |  |  |  | 1.13 (0.175)
  2 years to <6 years (n=0, 0, 0, 0, 0, 0, 7) |  | NA (NA) — Not assessed |  |  |  |  | 1.05 (0.089)
  6 years to <12 years (n=0, 0, 0, 0, 0, 0, 8) |  | NA (NA) — Not assessed |  |  |  |  | 1.04 (0.088)
  12 years to 17 years (n=0, 11, 0, 0, 0, 0, 0) |  | 0.614 (0.251) |  |  |  |  | NA (NA) — Not assessed

7. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product. Participants were monitored for the occurrence AEs for up to 14 days after last dose of study drug.
Time Frame: Up to 14 days after last dose of study drug (Up to 17 days)
Population: The All Subjects as Treated (ASaT) population consisted of all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Part IA-fosaprepitant 115 mg/Aprepitant | Part IB-fosaprepitant 150 mg | Part IIA-aprepitant 80 mg Equiv. | Part IIB-aprepitant 125 mg Equiv. | Part III-ondansetron | Part IV-aprepitant Regimen | Part V-fosaprepitant Regimen
Number analyzed (Participants) | 12 | 11 | 19 | 19 | 19 | 20 | 23
Participants | 11 | 6 | 18 | 16 | 15 | 13 | 17

8. Secondary Outcome: Plasma Concentration and PK Parameters of Dexamethasone in Participants From Birth to 1 Year of Age
Description: Blood samples for PK assessment were to be collected at the following time points: Parts II and V - Pre-dose and 1.5, 3, 4, 6, 8 and 24 hr post start of chemotherapy; Parts III and IV - Immediately after infusion of dexamethsone and 0.5, 1.5, 3, 8 and 24 hr post start of chemotherapy.
Time Frame: Up to 24 hours post dexamethasone dose
Population: This population was to consist of all participants from birth to 1 year of age who received at least one dose of dexamethasone and were evaluable for this PK parameter. These analyses were not conducted; enrollment of this cohort was not opened as enrollment of participants from birth to <6 months of age into Part II was unsuccessful.
Arm/Group | Part IA-fosaprepitant 115 mg/Aprepitant | Part IB-fosaprepitant 150 mg | Part IIA-aprepitant 80 mg Equiv. | Part IIB-aprepitant 125 mg Equiv. | Part III-ondansetron | Part IV-aprepitant Regimen | Part V-fosaprepitant Regimen
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants Discontinuing Study Drug Due to an AE
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product. The number of participants who discontinued from the study due to an AE are summarized.
Time Frame: Day 1 up to Day 3
Population: The ASaT population consisted of all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Part IA-fosaprepitant 115 mg/Aprepitant | Part IB-fosaprepitant 150 mg | Part IIA-aprepitant 80 mg Equiv. | Part IIB-aprepitant 125 mg Equiv. | Part III-ondansetron | Part IV-aprepitant Regimen | Part V-fosaprepitant Regimen
Number analyzed (Participants) | 12 | 11 | 19 | 19 | 19 | 20 | 23
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 14 days after last dose of study drug (Up to 17 days)
Description: The ASaT population consisted of all randomized participants who received at least one dose of study drug. Participants who completed Part III could enter Parts IV and V, and are counted once for each study part in which they participated. AEs are reported based on the study drug taken at the time of the event.
Arm/Group | Part IA-fosaprepitant 115 mg/Aprepitant | Part IB-fosaprepitant 150 mg | Part IIA-aprepitant 80 mg Equiv. | Part IIB-aprepitant 125 mg Equiv. | Part III-ondansetron | Part IV-aprepitant Regimen | Part V-fosaprepitant Regimen
Serious Adverse Events (participants affected / at risk) | 4/12 | 1/11 | 7/19 | 4/19 | 5/19 | 2/20 | 9/23
Other Adverse Events (participants affected / at risk) | 11/12 | 5/11 | 18/19 | 15/19 | 15/19 | 13/20 | 16/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part IA-fosaprepitant 115 mg/Aprepitant (N=12) | Part IB-fosaprepitant 150 mg (N=11) | Part IIA-aprepitant 80 mg Equiv. (N=19) | Part IIB-aprepitant 125 mg Equiv. (N=19) | Part III-ondansetron (N=19) | Part IV-aprepitant Regimen (N=20) | Part V-fosaprepitant Regimen (N=23)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 4 (4) | 2 (2) | 4 (4) | 2 (2) | 4 (4)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulval abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part IA-fosaprepitant 115 mg/Aprepitant (N=12) | Part IB-fosaprepitant 150 mg (N=11) | Part IIA-aprepitant 80 mg Equiv. (N=19) | Part IIB-aprepitant 125 mg Equiv. (N=19) | Part III-ondansetron (N=19) | Part IV-aprepitant Regimen (N=20) | Part V-fosaprepitant Regimen (N=23)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 5 (5) | 5 (5) | 3 (3) | 3 (3)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 3 (3) | 3 (3) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 4 (5) | 5 (5) | 4 (5)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 1 (1) | 3 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0) | 2 (3) | 6 (6) | 0 (0) | 1 (2) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Perianal erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (7) | 0 (0) | 9 (23) | 8 (21) | 2 (2) | 1 (1) | 5 (7)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Implant site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritability (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Product taste abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 7 (8)
Secretion discharge (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Oral bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotranferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug clearance decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glucose urine present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Formication (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Perineal erythema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.